CLINICAL TRIAL: NCT04245904
Title: Comparison of Respiratory Functions and Physical Fitness Parameters of Professional Basketball Players With Sedentary Controls
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Hilal GÜNGÖR, Comparison of Respiratory Functions and Physical Fitness Parameters of Professional Basketball Players with Sedentary Controls, Hacettepe University
Other Study IDs: GO 19/52
Record Dates: First submitted 2019-12-28; First posted 2020-01-29 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Physical Fitness, Basketball, Respiratory
Keywords: basketball, respiratory, physical fitness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- proffesional basketball player
- sedentary control

SUMMARY:
The aim of the study was to compare the professional basketball players and sedentary controls in terms of respiratory function and physical fitness parameters and to investigate the relationship between respiratory function and physical fitness parameters in basketball players.

DETAILED DESCRIPTION:
Basketball is one of the most common team sports in the world, where aerobic and anaerobic power is used together and taking into account the rising number of participants in non-professional leagues, it is especially popular among female athletes from various countries . Basketball players' muscular strength and endurance, power, speed, agility and physical properties such as reaction time are the main factors underlying the performance. In addition to this, respiratory functions are important as well as physical properties in basketball. Because during the maximal exercise, the blood flow to the inspiratory and expiratory muscles accounts for 15% of the total oxygen cost of the exercise. Assessment of the motor skills and physical characteristics of basketball players is very important for the positioning of the player, performance analysis and monitoring the effectiveness of the training. There are many studies examining the physical fitness characteristics of basketball players.However, no study evaluating respiratory muscle strength and endurance in female basketball players was found in the literature.therefore, this study was planned.

ELIGIBILITY:
Inclusion Criteria:

-

Inclusion criteria of basketball players:

* Female athletes with at least 3 years of professional basketball experience
* Volunteer to participate in the study
* 18-35 years
* Participating in training sessions regularly
* Non-smoking
* Do not use any supplements or medicines that affect physical performance

The inclusion criteria for healthy sedentaries were:

* 18-35 years old women
* Volunteering
* Have never done sports
* No smoking

Exclusion Criteria:

* • Doing any sport except basketball

  * Chronic respiratory or cardiovascular disease
  * Have had respiratory tract infection at least 4 weeks before the test (potential effect on respiratory muscle strength)
  * Have had an orthopedic injury in the last 3 months
  * Abandoned tests for any reason
  * Leaving the team or transferring to another team

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A team playing professional basketball in Turkey in Super League Basketball Women Study (mean age, 24.24 ± 4.96 years), basketball and sedentary individuals of the same age and sex were included on a voluntary basis. Permits were obtained from the necessary institutions before the studies to be made to the athletes. A total of 42 people from 21 people were included in the study according to 5% Type1 error, two-way hypothesis test design and sample size calculation with at least 80% working power. Before the measurement protocols, the participants were informed about the study and informed consent form was obtained.
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-06-08 (Actual)

PRIMARY OUTCOMES:
respiratory muscle strenght | day 1
  Respiratory muscle strength was assessed by an electronic mouth pressure measuring device (Micro Medical, Kent, UK) measuring MIP and MEP according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria . At least three measurements were taken. Between the measurements were given 1 minute rest. MIP was measured during deep inspiration after expiration up to the residual volume. Nasal respiration was prevented with the help of clips by asking the participants to evacuate all air from the nose and they were asked to breathe with maximum inspiratory effort. MEP was measured during deep expiration up to total lung capacity. After nasal breathing was prevented, the person was asked to exhale with maximum effort . Values were calculated according to age and gender variables using Black and Haytt's reference thresholds and recorded as a percentage of expected values.
respiratory muscle endurance | day 1
  Respiratory muscle endurance was measured by the incremental load testing with Power Breathe (HaB International Ltd. Southam, UK). The test was completed when it was not tolerated in case of shortness of breath and fatigue. The duration of the person's performance in different workloads was recorded. A workload level of less than one minute is considered invalid and a lower level is recorded. The results are obtained by multiplying the maximum workload in more than one minute and time values in seconds.
Total body weight | day 1
  Total body weight (kg) of the participants were measured using a digital scale (BC-418 MA, Tanita®, Japan) sensitive to fasting up to 0.1 kg on an empty stomach.
Body fat percentage | day 1
  Body fat percentage (%), of the participants were measured using a digital scale (BC-418 MA, Tanita®, Japan) sensitive to fasting up to 0.1 kg on an empty stomach.
fat free mass (FFM) | day 1
  (FFM) (kg) of the participants were measured using a digital scale (BC-418 MA, Tanita®, Japan) sensitive to fasting up to 0.1 kg on an empty stomach.
Body mass index | day 1
  The body mass index (BMI) of the participants was calculated according to the body weight / height2 (kg / m2) formula according to WHO criteria.
VO2max | day 2
  20 meters shuttle running test: It is a multistage test, commonly used to estimate VO2max, with the first stage being warming up. In this test, individuals performed 2X20 meter shuttle runs between the start and finish lines at a starting speed of 8.5 km / h and incremental speeds of 0.5 km / h per minute. The running speed was determined by automatic warning sounds from the CD player. The test consists of 21 levels and each level lasts 1 minute. The test was terminated when the participant ran out of power or delayed reaching the finish line twice. According to the score form of the test, the level of the participants' running was recorded and the "distance koş considered as the basis for the performance. VO2max total calculated distance was calculated by substituting in the formula (66.88).
  VO2max = 20.6 + Final stage completed x3 (88)
T-Drill test | day 2
  T-Drill Test for Agility The T-Drill test was performed using the protocol specified by Semenick (89). The three funnels were placed in the same direction with 5 yards (5 yards = 4.57 m) apart. The other funnel was placed at a distance of 10 yards from the center of the funnels (in the form of the letter T). It includes 5 steps to the left (5 yards = 4.57 m), 10 steps to the right (10 yards = 9.14 m), 5 steps to the left, 10 steps backwards. At the starting point (0 meters), the person finished the test with one of the knees in front and one in the back, then stepping forward, left, right, and backward at maximum speed. Three replicates were taken for each participant. 3 minutes of rest was given between each trial. The measurement results were recorded in seconds. The best score was used for statistical analysis after three trials (90).
20 m speed test | day 1
  The 20 meter (m) speed test was used for the speed values of the participants. Stopwatch was used for 20 m speed test. For the test, two cones at 20 m intervals and three cones in the form of a cone at 25 m were placed in the same direction. Participants were asked to continue up to 25 m so that they did not slow down without completing the test. The starting position of the participant was to place one of his feet not to exceed the exit funnel. The time until the person crossed the cone at 20 m was recorded after the person exited with the signal given while the participant was ready in the starting position. The test was taken 3 times at 2 min intervals. The values were saved in seconds. The shortest time was evaluated.
reaction time | day 2
  The reaction time was measured by Fitlight Trainer ™ (Fitlight Traniner Corperation, Thensvej, Risskov, Denmark). Hand reaction speed test: With the Fitlight TrainerTM, six LED lights placed at certain points on the wall were lit randomly and the person was asked to turn them off as fast as possible. In the protocol, the LEDs were placed according to the physical structure of the person and the number of seconds in which the 29 LEDs were extinguished were recorded in seconds .

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No